CLINICAL TRIAL: NCT01721512
Title: The Growth and Development of Breast and Formula Fed (Containing Synbiotics and LCPUFA) Term Asian Infants.
Brief Title: The Growth and Development of Breast and Formula Fed Term Asian Infants
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: Fonterra Brands (Singapore) PTE LTD (Unknown)
Responsible Party: Principal Investigator, Prof. Agus Firmansyah, MD, Ph.D, Professor and Chief, Division of Gastrohepatology, Department of Child Health, Medical Faculty, University of Indonesia, Indonesia University
Other Study IDs: Project Grow
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Growth
Keywords: Prospective observational study; Breast feeding; Infant formula; Infant; Indonesia
MeSH Terms: conditions — Breast Feeding | interventions — Lactation; Infant Formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast-fed infants: 80 infants of mothers who plan to exclusively breastfeed for at least 6 months.
  Interventions: Other: Breastfeeding
- Formula-fed infants: 1. Mother is exclusively feeding infant formula milk less than or equal to 6 weeks of birth and has no prospect of breastfeeding.
  2. Mother consents to her infant receiving trial infant formula for 12 months
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Breastfeeding
  Groups: Breast-fed infants
Other: Infant formula
  Groups: Formula-fed infants

SUMMARY:
Prospective cohort study of breast and formula fed infants in a suburban setting in Jakarta, Indonesia

ELIGIBILITY:
Inclusion Criteria:

* Breast-fed: 1. Mother intends to exclusively breast-feed from birth to at least 4 months; 2. A healthy term infant with gestational age fo 37-42 weeks and birth weight greater than or equal to 2.5 kg and equal or less than 4.75 kg.
* Formula-fed: 1. Mother is exclusively feeding infant formula milk less than or equal to 6 weeks of birth and has no prospect of breastfeeding; 2. A healthy term infant with gestational age fo 37-42 weeks and birth weight greater than or equal to 2.5 kg and equal or less than 4.75 kg; 3. Mother consents to her infant receiving trial infant formula for 12 months.

Exclusion Criteria:

* 1. Severe congenital or metabolic disease likely to affect infant feeding or infant growth.
* 2. Multiple birth

Ages: 2 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants recruited from Jati Padang, Pasar Minggu District, South Jakarta, Indonesia
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Infant weight, body length head circumference | 12 months
  Infant weight, body length head circumference at enrolment, 2 weeks, 4 weeks and monthly thereafter until 6 months, and then at 8, 10 and 12 months.

SECONDARY OUTCOMES:
Gastrointestinal tolerance | 6 months
  Gastrointestinal tolerance: stool frequency and consistency using Bristol Stool Chart monthly up to 6 months
Indicators or formula tolerance | 12 months
  Indicators or formula tolerance: crying, irritability, sleep patterns
General health | 12 months
  General health: any hospitalisation, doctor visits, symptoms of respiratory or gastrointestinal infection, fever, antibiotic and medication usage
Gut integrity | 3 months
  Gut integrity: faecal Alpha1-antitrypsin and faecal calprotectin
Gut microflora | 3 months
  Gut microflora: real time PCR
Developmental progress | 12 months
  Developmental progress: assessed by Ages and Stages

CONTACTS AND LOCATIONS:
Overall Officials: Agus Firmansyah, Professor, MD, PhD, SpA(K), Principal Investigator — Indonesia University
Locations (1):
- Universitas Indonesia, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Derived] Dwipoerwantoro PG, Mansyur M, Oswari H, Makrides M, Cleghorn G, Firmansyah A. Growth of Indonesian Infants Compared With World Health Organization Growth Standards. J Pediatr Gastroenterol Nutr. 2015 Aug;61(2):248-52. doi: 10.1097/MPG.0000000000000770. PMID 25710823